CLINICAL TRIAL: NCT04216277
Title: The Procalcitonin Guided Antibiotics in Respiratory Infections in General Practice
Acronym: PARI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the poc test was withdrawn by manufacturer
Sponsor: Chronic Obstructive Pulmonary Disease Trial Network, Denmark (Other)
Collaborators: Research Unit Of General Practice, Copenhagen (Other); Department of Public Health, Denmark (Other)
Responsible Party: Principal Investigator, Rune Munck Aabenhus, MD. Specialist in General Practice, PhD, Assistent Professor, Chronic Obstructive Pulmonary Disease Trial Network, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18057336
Record Dates: First submitted 2019-12-12; First posted 2020-01-02 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Tract Infection
Keywords: primary care; acute respiratory tract infection; Procalcitonin; general practice; Antibiotic use

STUDY DESIGN:
Who Masked: Participant
Masking Description: Procalcitonin will be measured on all participants but none of the participants will be informed about the results of the procalcitonin value or the randomisation and thus remain unaware of allocated group status (intervention or control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Procalcitonin in addition to usual care (Experimental): Procalcitonin values will be disclosed to the attending physician and assist in antibiotic guidance in addition to usual care
  Interventions: Diagnostic Test: Procalcitonin
- Usual care (No Intervention): Usual best standard care. No procalcitonin values disclosed to attending physician .

INTERVENTIONS:
Diagnostic Test: Procalcitonin — In addition to usual care diagnostic and handling of acute respiratory tract infections in general practice to attending physician in the intervention arm has access to antibiotic stewardship by a procalcitonin point-of-care test. The following criteria for initiating og withholding antibiotics will be used.
  * Antibiotics treatment is recommended with Procalcitonin levels above 0.25 ng/ml
  * Antibiotic treatment is discouraged if Procalcitonin levels are below 0.25 ng/ml
  Arms: Procalcitonin in addition to usual care

SUMMARY:
Antimicrobial resistance rates have reached alarming levels and the Worlds Health Organisation (WHO) states it constitutes a serious public health concern by threatening one of the most effective and mortality lowering interventions in modern medicine. Part of the solution to this problem includes minimizing overuse of antibiotics. But clinical signs alone are often not reliable to guide antibiotic treatment decisions and additional tests may be warranted to assist the doctor. Such tests include point-of-care biomarkers of infection like C-reactive protein (CRP) and procalcitonin (PCT). Targeting antibiotic use to the few patients with a high probability of benefit and withholding in the many with non-serious respiratory infection is a promising strategy and readily implemented in clinical practice.

The Procalcitonin guided Antibiotics in Respiratory Infections (PARI) study will assess the effect of a novel point-of-care PCT guided antibiotic stewardship in acute respiratory tract infections in general practice.

The overall aim of the PARI study is to reduce antibiotic use in patients with acute respiratory tract infections by targeting antibiotic treatment only to patients with a suspected bacterial etiology and thus likely to benefit from antibiotic therapy.

The main research questions are:

Does the addition of a point-of-care Procalcitonin test to standard care reduce antibiotic use in primary care? Is the intervention safe for the patients? The PARI study is a pragmatic two-arm (intervention and control (standard care) open randomized non-inferiority trial (up to 1 day difference in recovery) in general practice.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Able to read and understand patient information about the PARI trial and willing to give written informed consent prior to enrollment
* Acute cough e.g. less than 2 weeks probable acute upper or lower respiratory tract infection (pharyngitis, tonsillitis, otitis media, sinusitis, exacerbations of asthma or Chronic Obstructive Pulmonary Disease (COPD), bronchitis or pneumonia)
* C-Reactive Protein >20 mg/m

Exclusion Criteria:

* Symptoms present for more than 2 weeks
* Verified immunodeficiency or presently neutropenic (neutrophile granulocytes ≤0,5 x 109/L within the last 7 days)
* Severe liver failure
* Severe kidney failure including dialysis
* Sore throat and positive test for Group A streptococcus
* Prior antibiotic exposure last 14 days up to inclusion
* Need for acute admission to hospital
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Duration of illness and symptoms from acute respiratory tract infections. | up to 14 days
  The patient reported primary outcome will be assessed as number of days to a patient's daily activities (work or recreation) are no longer restricted by symptoms from a respiratory tract infection.The non-inferiority margin between the intervention and control group is set at a one day difference. The recovery measure will be the specific day indicated by the participants using the validated Acute Respiratory Tract Infections Questionaire (ARTIQ).

SECONDARY OUTCOMES:
Antibiotic treatments | 1, 14 and 30 days
  Number of participants in each trial arm exposed to antibiotic treatment at index consultation (day 1) and within 30 days
Side effects from antibiotic treatment | 14 days
  Number of participants in each trial arm with side effects from antibiotic treatment
re-consultations | 30 days
  Number of participants in each trial arm with re-consultations
Severe adverse effects | 30 days
  Number of participants in each trial arm admitted to hospitalization (including diagnosis and mortality)
Biomarker levels | day 1
  Characterisation of biomarker (C-Reactive Protein and Procalcionin) levels at index consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjerrum, PhD, Study Chair — Department of Public Health, Copenhagen University, Denmark
Locations (6):
- Denmark (6):
  - Lægerne Finne, Riise og Aabenhus, Copenhagen
  - Amagercentrets læger, Copenhagen
  - Mit Lægehus, Copenhagen
  - Haslev Lægecenter, Haslev
  - Næstved Lægecenter, Næstved
  - Rønnede lægehus, Rønnede

IPD SHARING:
Plan to Share IPD: Yes
work in progress
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon publication of study results

REFERENCES:
- [Derived] Filipsen N, Bro H, Bjerrum L, Jensen JS, Aabenhus R. The Procalcitonin-guided Antibiotics in Respiratory Infections (PARI) project in general practice - a study protocol. BMC Prim Care. 2022 Mar 12;23(1):43. doi: 10.1186/s12875-022-01646-6. PMID 35279069